CLINICAL TRIAL: NCT05889637
Title: Gastric Ultrasound Assessment for Preoperative Prandial State of Patients Taking Glucagon-Like Peptide-1(GLP-1) Receptor Agonists
Brief Title: Gastric Ultrasound Assessment for Preoperative Prandial State of Patients Taking Glucagon-Like Peptide-1 Receptor Agonists
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sudipta Sen, Assisstant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-23-0300
Record Dates: First submitted 2023-05-08; First posted 2023-06-05 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group G: Patients taking GLP-1receptor agonists
  Interventions: Diagnostic Test: Gastric ultrasound
- Group C: Patients not taking GLP-1 receptor agonists (control group)
  Interventions: Diagnostic Test: Gastric ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric ultrasound — Patient will be scanned first in the supine position and then in the right lateral decubitus position. The ultrasound probe will be placed in a sagittal plane in the epigastric region at the left subcostal margin and then will be moved past the midline in a fan like manner to the right subcostal region. Qualitative and quantitative assessments will be done.

SUMMARY:
The purpose of this study is to determine the type of gastric content and quantify the volume of liquid gastric contents using ultrasonography in patients on GLP-1 agonists that have presented for elective surgery and to determine if risk factors are associated with a higher gastric volume in patients on GLP-1 receptor agonists.

ELIGIBILITY:
Inclusion Criteria:

* Patients taking GLP-1receptor agonists (N=62)
* Patients not taking GLP-1 receptor agonists (N=62)

Exclusion Criteria:

* Previous gastric resection or bypass
* Gastric band in situ
* Previous fundoplication
* Large hiatal hernia
* Pregnant patients
* Recent trauma
* Inability to turn to the right lateral decubitus position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects presenting for elective surgery who are on Glucagon-Like peptide-1 agonist subcutaneous injection, once weekly will be included
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects that are at risk for aspiration | end of ultrasound
  Risk for aspiration is indicated by the presence of solids, thick fluid, or clear fluids >1.5ml/kg in the gastric antrum in the right lateral decubitus position
Number of subjects that are at low risk for aspiration | end of ultrasound
  Low risk for aspiration is indicated by a collapsed gastric antrum or clear fluids <1.5ml/kg in the gastric antrum in the right lateral decubitus position.

SECONDARY OUTCOMES:
Age | end of ultrasound
Number of participants that are male as indicated in the medical records | end of ultrasound
Number of participants that are female as indicated in the medical records | end of ultrasound
Body mass Index (BMI) | end of ultrasound
  Body Mass Index (BMI) is calculated as the body mass in kilograms (kg) divided by the square of the body height in meters, and is expressed in units of kg/m2.
Physical status as assessed by the American Society of Anesthesiologists (ASA) physical status classification system | end of ultrasound
  The classification ranges from American Society of Anesthesiologists (ASA)1 (normal healthy person ) to ASA IV (A patient with severe systemic disease that is a constant threat to life)
Number of participants with diabetes | end of ultrasound
Number of participants with reported nothing by mouth (NPO) status | end of ultrasound
Pain severity as assessed by the numeric scale | end of ultrasound
  This is a 11 point scale with scores ranging from 0 (no pain) to 10 (worst imaginable pain)
Number of participants with Gastroesophageal reflux disease (GERD) | end of ultrasound
Number of participants that have use opioids preoperatively | end of ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Sudipta Sen, MD,FASA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No